CLINICAL TRIAL: NCT04745949
Title: A Phase II Study to Determine the Response Kinetics, Safety, and Efficacy of Brentuximab Vedotin and Nivolumab Alone and Then Combined With Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone for Patients With Untreated Primary Mediastinal Large B-Cell Lymphoma
Brief Title: PACIFIC: Primary Mediastinal Large B-cell Lymphoma Treated With Antibody Therapy, Checkpoint Inhibitor in Frontline With ImmunoChemotherapy
Acronym: PACIFIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0686; NCI-2020-13888 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0686 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Ann Arbor Stage I Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Ann Arbor Stage II Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Ann Arbor Stage III Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Ann Arbor Stage IV Primary Mediastinal (Thymic) Large B-Cell Lymphoma
Keywords: Primary Mediastinal Large B-cell Lymphoma; Brentuximab Vedotin; Nivolumab; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone
MeSH Terms: interventions — Brentuximab Vedotin; Cyclophosphamide; Doxorubicin; Nivolumab; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (brentuximab vedotin, nivolumab, R-CHP) (Experimental): Patient will receive an immune lead-in of 2 cycles of Brentuximab vedotin and Nivolumab (A-O) (cycles 1 and 2), which has an appropriate futility rules in place to close early if efficacy targets are not met. At cycle 3 and 4, patients will receive A-O with R-CHP. Patients who will have achieved complete response (CR) at PET/CT before cycle 5 will receive 2 more cycles of A-O-R-CHP (cycle 5 and 6) and A-O only for cycle 7 and 8. If these patients still present CR at PET/CT after cycle 8, they will have completed therapy and will be followed up. In case of stable disease or progressive disease at PET/CT after cycle 4, the patient will be taken off the trial. Patients who present further response but no CR, at PET/CT before cycle 5 will receive 4 more cycles A-O-R-CHP (cycles 5-8). If they reach CR at PET/CT after cycle 8, they will have completed therapy and will be followed up. All patients will receive a total of 8 cycles of A-O. The cycle duration is 21 days.
  Interventions: Drug: Brentuximab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Nivolumab; Drug: Prednisone; Other: Quality-of-Life Assessment; Biological: Rituximab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies the effect of brentuximab vedotin and nivolumab alone and in combination with rituximab, cyclophosphamide, doxorubicin, and prednisone in treating patients with untreated, stage I-IV primary mediastinal large B-cell lymphoma. Brentuximab vedotin is a monoclonal antibody, called brentuximab, linked to a toxic agent, called vedotin. Brentuximab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD30 receptors, and delivers vedotin to kill them. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Rituximab is a type of antibody therapy, which targets and attaches to the CD20 protein found on the surface of blood cells with cancer and some healthy blood cells. Chemotherapy drugs, such as cyclophosphamide, and doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, or by stopping them from dividing. Prednisone is a steroid, a hormone (chemical messengers) with multiple roles, notably in the immune system and inflammation reduction. Steroids are poisonous to lymphocytes (white blood cells from which lymphomas develop). Giving brentuximab vedotin and nivolumab in combination with rituximab, cyclophosphamide, doxorubicin, and prednisone may help to control the disease and be a less harmful regimen than standard chemotherapy in patients with primary mediastinal large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of primary mediastinal large B-cell lymphoma (PMBL) patients treated brentuximab vedotin (A) and nivolumab (O) alone and then combined with rituximab, cyclophosphamide, doxorubicin, and prednisone (R-CHP).

SECONDARY OBJECTIVE:

I. Evaluate the antitumor activity, safety, tolerability, patient reported quality of life and survival of brentuximab vedotin and nivolumab (A-O) alone and then combined with R-CHP in patients with untreated PMBL.

EXPLORATORY OBJECTIVE:

I. To evaluate the baseline and therapy induced changes in the profile of mutations and gene expression.

OUTLINE:

Patient will receive an immune lead-in of 2 cycles of Brentuximab vedotin and Nivolumab (A-O) (cycles 1 and 2), which has an appropriate futility rules in place to close early if efficacy targets are not met. At cycle 3 and 4, patients will receive A-O with R-CHP. Patients who will have achieved complete response (CR) at PET/CT before cycle 5 will receive 2 more cycles of A-O-R-CHP (cycle 5 and 6) and A-O only for cycle 7 and 8. If these patients still present CR at PET/CT after cycle 8, they will have completed therapy and will be followed up. In case of stable disease or progressive disease at PET/CT after cycle 4, the patient will be taken off the trial. Patients who present further response but no CR, at PET/CT before cycle 5 will receive 4 more cycles A-O-R-CHP (cycles 5-8). If they reach CR at PET/CT after cycle 8, they will have completed therapy and will be followed up. All patients will receive a total of 8 cycles of A-O. The cycle duration is 21 days. Brentuximab vedotin will be given intravenously (IV) over 30 minutes and nivolumab IV over 30 minutes on day 1. R-CHP: rituximab IV will be administered over 4-6 hours, cyclophosphamide IV over 1 hour, and doxorubicin IV over 1 hour on day 1, and prednisone orally (PO) once daily (QD) on days 1-5.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of PMBL

  * Require a CD30 expression level of 1% or greater in the tumor or tumor-infiltrating lymphocytes by local immunohistochemistry
* No prior treatment except

  * A prior limited-field radiotherapy
  * A short course (up to 7 days) of glucocorticoids =< 100 mg daily of prednisone equivalent which must cease prior to day 1 of cycle 1
* Stage of patients: Stages II, III, IV, and stage I >= 5 cm in the greatest dimension
* Patient or durable power of attorney (DPA) for healthcare must be able to understand and voluntarily sign an Institutional Review Board (IRB)-approved informed consent form
* Age >= 18 years at the time of signing the informed consent
* Patients must have bi-dimensional measurable disease, as defined as radiographically apparent disease with the longest dimension of >= 1.5 cm
* Patients with performance status of =< 3 (3 only allowed if decline in status is deemed related to lymphoma and felt potentially reversible by the treating physician)
* Serum bilirubin < 1.5 x ULN except in patients with Gilbert's syndrome as defined by > 80% unconjugated bilirubin
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN or < 5 x ULN if hepatic metastases are present
* Absolute neutrophil count (ANC) > 1000/mm^3 unless deemed related to lymphoma involvement in the bone marrow and felt potentially reversible by the treating physician
* Platelets > 1000/mm^3 unless deemed related to lymphoma involvement in the bone marrow and felt potentially reversible by the treating physician
* Calculated creatinine clearance >= 30 ml/min by Cockcroft-Gault formula
* Patients must be willing to receive transfusions of blood products
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at screening
* Women of childbearing potential and men who are sexually active with a woman of childbearing potential must be practicing a highly effective method of birth control during and after the study (12 months for women and 3 months for men), consistent with local regulations regarding the use of birth control methods for subjects participating in this clinical study. Men must agree to not donate sperm during and for up to 3 months after their conclusion of therapy on study. For females, these restrictions apply for 1 month after the last dose of study drug

Exclusion Criteria:

* Patients with an urgent need for cytoreductive treatment will be excluded
* Any serious medical condition including but not limited to uncontrolled hypertension, uncontrolled congestive heart failure within past 6 months prior to screening (class 3 [moderate] or class 4 [severe] cardiac disease as defined by the New York Heart Association Functional Classification), uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), left ventricular ejection fraction (LVEF) less than 40%, renal failure, active infection, history of invasive fungal infection, moderate to severe hepatic disease (Child Pugh class B or C), active hemorrhage, laboratory abnormality, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form. Patients with history of cardiac arrhythmias should have cardiac evaluation and clearance
* Previous anthracycline exposure with expected lifetime exposure to doxorubicin > 450 mg/m^2, considering the planned anthracycline exposure in this study with potential six cycles of R-CHP
* Pregnant or lactating females
* Known hypersensitivity to brentuximab vedotin, nivolumab, rituximab, doxorubicin, cyclophosphamide, or prednisone
* Known human immunodeficiency virus (HIV) infection with active viremia

  * Patient with known HIV infection can be included if undetectable viral load, CD4 >= 300 cells/microL and on HAART (highly active antiretroviral therapy)
* Patients with active viremia of hepatitis B infection

  * Not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody
* Patients with active viremia of hepatitis C infection

  * Known hepatitis C infection is allowed as long as there is no active disease and is cleared by gastrointestinal (GI) consultation
* All patients with central nervous system involvement with lymphoma
* Diagnosis of prior malignancy within the past 2 years with the exception of successfully treated basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast. History of other malignancies are allowed if in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years
* Significant neuropathy (grades 2 or grade 1 with pain) within 14 days prior to enrollment
* Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis not due to lymphoma
* Major surgery within 4 weeks of study entry or wound that is not healed from prior surgery or trauma
* History of stroke or intracranial hemorrhage within 6 months prior to study entry
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2027-08-03 (Estimated); Study Completion 2027-08-03 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At completion of therapy, assessed up to 2 years
  Will be defined as the percentage of number of complete responses in total number of patients treated, which includes all the patients who were treated, even the patients dropped out at interim positron emission tomography/computed tomography scan after cycle 4 due to stable disease/progressive disease. Simon's optimal two-stage design will be used. Fisher's exact test will be used to evaluate the association between response and other categorical patient variables. T-test or Wilcoxon rank sum test will be used to evaluate the difference in continuous variables between responders and non-responders.

SECONDARY OUTCOMES:
Overall response rate (complete response + partial response) | Up to 2 cycles of brentuximab vedotin and nivolumab (1 cycle = 21 days)
  Will monitor the overall response using the Bayesian stopping boundaries calculated based on beta-binomial distributions, and 95% confidence intervals will be calculated. Fisher's exact test will be used to evaluate the association between response and other categorical patient variables. T-test or Wilcoxon rank sum test will be used to evaluate the difference in continuous variables between responders and non-responders.
1-year progression-free survival | From study entry to objective disease progression or death from any cause, whichever occurs first, assessed at 1 year
  Will be estimated using the method of Kaplan and Meier.
2 -year progression-free survival | From study entry to objective disease progression or death from any cause, whichever occurs first, assessed at 2 years
  Will be estimated using the method of Kaplan and Meier.
1-year overall survival | From study entry to death from any cause, assessed at 1 year
  Will be estimated using the method of Kaplan and Meier.
2-year overall survival | From study entry to death from any cause, assessed at 2 years
  Will be estimated using the method of Kaplan and Meier.
Duration of response | Up to 2 years post-treatment
Incidence of adverse events | Up to 100 days of the last dose of the study drug
  Will be summarized by frequency tables for all patients.
Health-related quality of life | Up to 2 years post-treatment
  Will be assessed by the European Organization of Research and Treatment of Cancer Quality of Life Questionnaire - Core (C) 30 (EORTC QLQ-C30).

OTHER OUTCOMES:
Minimal residual disease clonotype levels | Up to 2 years post-treatment
  Will be assessed in tumor biopsy and blood samples.
Cell free deoxyribonucleic acid | Up to 2 years post-treatment
  Will be assessed in tumor biopsy and blood samples.
Immune cell subsets | Up to 2 years post-treatment
  Will be assessed in tumor biopsy and blood samples.
Tumor protein expression | Up to 2 years post-treatment
  Will be assessed in tumor biopsy and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Nair, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org